## Investigational device exemption G010002 Endovascular Exclusion of TAAA or AAA utilizing Fenestrated or Branched Data analysis plan for annual FDA report

Written: 7 December 2005 Last modified: 9 March 2006

### 1. Definitions of image-related events

At each follow-up imaging visit (each value of FIMG:CPEVENT), each patient is classified as follows:

endoleak, any

| yes if | on follow-up fenestrated imaging form,<br>endoleak = yes (FIMG:ENDOYN = |
|---|---|
| | "YES") |
| no if | on follow-up fenestrated imaging form, |
| | endoleak = no (FIMG:ENDOYN = "NO") |
| missing otherwise | |

endoleak, type I

| yes if | on follow-up fenestrated imaging form, |
|-------------------|----------------------------------------|
| | type I is checked (FIMG:ENDTYP1 = 1) |
| no if | on follow-up fenestrated imaging form, |
| | endoleak has been answered |
| | (FIMG:ENDOYN = "YES" or |
| | FIMG:ENDOYN = "NO") AND |
| | on follow-up fenestrated imaging form, |
| | type I is not checked (FIMG:ENDTYP1 = |
| | NULL) |
| missing otherwise | |

endoleak, type II

| endoreak, type n | |
|-------------------|----------------------------------------|
| yes if | on follow-up fenestrated imaging form, |
| | type II is checked (FIMG:ENDTYP2 = 1) |
| no if | on follow-up fenestrated imaging form, |
| | endoleak has been answered |
| | (FIMG:ENDOYN = "YES" or |
| | FIMG:ENDOYN = "NO") AND |
| | on follow-up fenestrated imaging form, |
| | type II is not checked (FIMG:ENDTYP2 = |
| | NULL) |
| missing otherwise | |

endoleak, type III

| yes if | on follow-up fenestrated imaging form,<br>type III is checked (FIMG:ENDTYP3 = 1) |
|---|---|
| no if | on follow-up fenestrated imaging form,<br>endoleak has been answered<br>(FIMG:ENDOYN = "YES" or<br>FIMG:ENDOYN = "NO") AND |
| | on follow-up fenestrated imaging form,<br>type III is not checked (FIMG:ENDTYP3<br>= NULL) |
| missing otherwise | |

endoleak, type IV

| endoreak, type 1 v | |
|--------------------|----------------------------------------|
| yes if | on follow-up fenestrated imaging form, |
| | type IV is checked (FIMG:ENDTYP4 = 1) |
| no if | on follow-up fenestrated imaging form, |
| | endoleak has been answered |
| | (FIMG:ENDOYN = "YES" or |
| | FIMG:ENDOYN = "NO") AND |
| | on follow-up fenestrated imaging form, |
| | type IV is not checked (FIMG:ENDTYP4 |
| | = NULL) |
| missing otherwise | |

endoleak, unknown

| yes if | on follow-up fenestrated imaging form,<br>unknown is checked (FIMG:ENDTYP5 =<br>1) |
|---|---|
| no if | on follow-up fenestrated imaging form,<br>endoleak has been answered<br>(FIMG:ENDOYN = "YES" or<br>FIMG:ENDOYN = "NO") AND |
| | on follow-up fenestrated imaging form,<br>unknown is not checked (FIMG:ENDTYP5<br>= NULL) |
| missing otherwise | |

# growth notation:

• A1\_p = maximum aneurysm diameter major axis on follow-up fenestrated imaging form (FIMG:DIAMEA1) at pre-discharge visit

- A1\_c = maximum aneurysm diameter major axis on follow-up fenestrated imaging form (FIMG:DIAMEA1) at current visit
- A2\_p = maximum aneurysm diameter minor axis on follow-up fenestrated imaging form (FIMG:DIAMEA2) at pre-discharge visit
- A2\_c = maximum aneurysm diameter minor axis on follow-up fenestrated imaging form (FIMG:DIAMEA2) at current visit

aneurysm growth (only defined for visits after pre-discharge [FIMG:CPEVENT = "PRE DISCHARGE"])

| yes if | A1 c - A1 p > 5 OR |
|-------------------|---------------------------------|
| | A2 c - A2 p > 5 |
| no if | $A1_c - A1_p \le 5 \text{ AND}$ |
| | $A2 c - A2 p \le 5$ |
| missing otherwise | |

aneurysm shrinkage (only defined for visits after pre-discharge [FIMG:CPEVENT = "PRE DISCHARGE"])

| yes if | $A1_c - A1_p < -5 OR$ |
|-------------------|----------------------------------|
| | $A2_c - A2_p < -5$ |
| no if | $A1_c - A1_p \ge -5 \text{ AND}$ |
| | $A2_c - A2_p \ge -5$ |
| missing otherwise | |

aneurysm stasis (only defined for visits after pre-discharge [FIMG:CPEVENT = "PRE DISCHARGE"])

| yes if | aneurysm growth = no AND |
|-------------------|--------------------------|
| | aneurysm shrinkage = no |
| no if | aneurysm growth = yes OR |
| | aneurysm shrinkage = yes |
| missing otherwise | |

#### migration notation:

- M4\_p = table position of uppermost proximal stent on follow-up fenestrated imaging form (FIMG:MIGTP4) at pre-discharge visit
- M4\_c = table position of uppermost proximal stent on follow-up fenestrated imaging form (FIMG: MIGTP4) at current visit
- M5\_p = table position of initial appearance of full circumference of stent on followup fenestrated imaging form (FIMG: MIGTP5) at pre-discharge visit
- M5\_c = table position of initial appearance of full circumference of stent on followup fenestrated imaging form (FIMG: MIGTP5) at current visit
- M1\_p = table position of SMA on follow-up fenestrated imaging form (FIMG: MIGTP1) at pre-discharge visit

• M1\_c = table position of SMA on follow-up fenestrated imaging form (FIMG: MIGTP1) at current visit

migration (only defined for visits after pre-discharge [FIMG:CPEVENT = "PRE\_DISCHARGE"])

| yes if | $ (M1_c - M4_c) - (M1_p - M4_p) > 10$ |
|-------------------|--------------------------------------------|
| | OR |
| | $ (M1_c - M5_c) - (M1_p - M5_p) > 10$ |
| no if | $ (M1_c - M4_c) - (M1_p - M4_p) \le 10$ |
| | AND |
| | $ (M1_c - M5_c) - (M1_p - M5_p) \le 10$ |
| missing otherwise | |

### stent fracture

| Stellt fracture | |
|---|---|
| yes if | on follow-up fenestrated KUB form,<br>proximal graft stent fracture = "YES"<br>(FKUB:DISF1 = "YES") OR |
| | on follow-up fenestrated KUB form, distal graft stent fracture = "YES" (FKUB:DISF2 = "YES") OR |
| | on follow-up fenestrated KUB form, right iliac stent fracture = "YES" (FKUB:DISF3 = "YES") OR |
| | on follow-up fenestrated KUB form, left iliac stent fracture = "YES" (FKUB:DISF4 = "YES") OR |
| | on follow-up fenestrated KUB form,<br>occluder stent fracture = "YES"<br>(FKUB:DISF5 = "YES") OR |
| | on follow-up fenestrated KUB form,<br>converter stent fracture = "YES"<br>(FKUB:DISF6 = "YES") OR |
| | on follow-up fenestrated KUB form, right iliac leg extension stent fracture = "YES" (FKUB:DISF7 = "YES") OR |
| | on follow-up fenestrated KUB form, left iliac leg extension stent fracture = "YES" (FKUB:DISF8 = "YES") OR |
| | on follow-up fenestrated KUB form, main<br>body extension stent fracture = "YES"<br>(FKUB:DISF9 = "YES") OR |
| | on follow-up fenestrated KUB form, renal<br>stent right stent fracture = "YES"<br>(FKUB:DISF10 = "YES") OR |
| | on follow-up fenestrated KUB form, renal |

| | (TIDO) |
|---|---|
| | stent left stent fracture = "YES" |
| | (FKUB:DISF11 = "YES") OR |
| | on follow-up fenestrated KUB form, other stent fracture = "YES" (FKUB:DISF12 = "YES") |
| no if | on follow-up fenestrated KUB form,<br>proximal graft stent fracture = "NO" or<br>"N/A" (FKUB:DISF1 = "NO" or "N/A")<br>AND |
| | on follow-up fenestrated KUB form, distal<br>graft stent fracture = "NO" or "N/A"<br>(FKUB:DISF2 = "NO" or "N/A") AND |
| | on follow-up fenestrated KUB form, right iliac stent fracture = "NO" or "N/A" (FKUB:DISF3 = "NO" or "N/A") AND |
| | on follow-up fenestrated KUB form, left iliac stent fracture = "NO" or "N/A" (FKUB:DISF4 = "NO" or "N/A") AND |
| | on follow-up fenestrated KUB form,<br>occluder stent fracture = "NO" or "N/A"<br>(FKUB:DISF5 = "NO" or "N/A") AND |
| | on follow-up fenestrated KUB form,<br>converter stent fracture = "NO" or "N/A"<br>(FKUB:DISF6 = "NO" or "N/A") AND |
| | on follow-up fenestrated KUB form, right iliac leg extension stent fracture = "NO" or "N/A" (FKUB:DISF7 = "NO" or "N/A") AND |
| | on follow-up fenestrated KUB form, left iliac leg extension stent fracture = "NO" or "N/A" (FKUB:DISF8 = "NO" or "N/A") AND |
| | on follow-up fenestrated KUB form, main<br>body extension stent fracture = "NO" or<br>"N/A" (FKUB:DISF9 = "NO" or "N/A")<br>AND |
| | on follow-up fenestrated KUB form, renal stent right stent fracture = "NO" or "N/A" (FKUB:DISF10 = "NO" or "N/A") AND |
| | on follow-up fenestrated KUB form, renal stent left stent fracture = "NO" or "N/A" (FKUB:DISF11 = "NO" or "N/A") AND |
| | on follow-up fenestrated KUB form, other stent fracture = "NO" or "N/A" (FKUB:DISF12 = "NO" or "N/A") |
| missing otherwise | |

## barb fracture

| yes if | on follow-up fenestrated KUB form, barb<br>bend is checked (FKUB:PFSNIN1 = 1) OR |
|---|---|
| | , |
| | on follow-up fenestrated KUB form, |
| | proximal stent separation is checked |
| | (FKUB:PFSNIN3 = 1) OR |
| | on follow-up fenestrated KUB form, barb |
| | separation is checked (FKUB:PFSNIN2 = |
| | 1) |
| no if | on follow-up fenestrated KUB form, barb |
| | bend is not checked (FKUB:PFSNIN1 = |
| | NULL) AND |
| | on follow-up fenestrated KUB form, |
| | proximal stent separation is not checked |
| | (FKUB:PFSNIN3 = NULL) AND |
| | on follow-up fenestrated KUB form, barb |
| | separation is not checked |
| | (FKUB:PFSNIN2 = NULL) |
| missing otherwise | |

component separation

| yes if | on follow-up fenestrated KUB form, "Has component separation of the endovascular graft occurred?" = "YES" |
|---|---|
| | (FKUB:COMSYN = "YES") |
| no if | on follow-up fenestrated KUB form, "Has component separation of the endovascular graft occurred?" = "NO" (FKUB:COMSYN = "NO") |
| missing otherwise | |

compression

| compression | |
|-------------|------------------------------------------|
| yes if | on follow-up fenestrated KUB form, renal |
| | stent right compression = "YES" |
| | (FKUB:DEVCPR1 = "YES") OR |
| | on follow-up fenestrated KUB form, renal |
| | stent left compression = "YES" |
| | (FKUB:DEVCPR2 = "YES") OR |
| | on follow-up fenestrated KUB form, other |
| | stent compression = "YES" |
| | (FKUB:DEVCPR3 = "YES") |
| no if | on follow-up fenestrated KUB form, renal |

| | stent right compression = "NO" or "N/A" (FKUB:DEVCPR1 = "NO" or "N/A") AND |
|---|---|
| | on follow-up fenestrated KUB form, renal<br>stent left compression = "NO" or "N/A"<br>(FKUB:DEVCPR2 = "NO" or "N/A")<br>AND |
| | on follow-up fenestrated KUB form, other stent compression = "NO" or "N/A" (FKUB:DEVCPR3 = "NO" or "N/A") |
| missing otherwise | |

occlusion, right iliac artery CIA

| yes if | on follow-up fenestrated imaging form, right iliac artery patent CIA = "YES" |
|---|---|
| | (FIMG:PATCIA1 = "NO") |
| no if | on follow-up fenestrated imaging form, right iliac artery patent CIA = "YES" (FIMG:PATCIA1 = "YES") |
| missing otherwise | |

occlusion, right iliac artery IIA

| yes if | on follow-up fenestrated imaging form, |
|-------------------|----------------------------------------|
| | right iliac artery patent IIA = "YES" |
| | (FIMG:PATIIA1 = "NO") |
| no if | on follow-up fenestrated imaging form, |
| | right iliac artery patent IIA = "YES" |
| | (FIMG:PATIIA1 = "YES") |
| missing otherwise | |

occlusion, left iliac artery CIA

| occiusion, ieit mac artery CIA | |
|--------------------------------|---------------------------------------------|
| yes if | on follow-up fenestrated imaging form, left |
| | iliac artery patent CIA = "YES" |
| | (FIMG:PATCIA2 = "NO") |
| no if | on follow-up fenestrated imaging form, left |
| | iliac artery patent CIA = "YES" |
| | (FIMG:PATCIA2 = "YES") |
| missing otherwise | |

occlusion, left iliac artery IIA

| yes if | on follow-up fenestrated imaging form, left |
|--------|---------------------------------------------|
| | iliac artery patent IIA = "YES" |

| | (FIMG:PATIIA2 = "NO") |
|-------------------|---------------------------------------------|
| no if | on follow-up fenestrated imaging form, left |
| | iliac artery patent IIA = "YES" |
| | (FIMG:PATIIA2 = "YES") |
| missing otherwise | |

occlusion, right renal

| _ coordston, right ronar | |
|--------------------------|----------------------------------------|
| yes if | on follow-up fenestrated imaging form, |
| | right renal occluded is checked |
| | (FIMG:PATRRA = "OCCLUDED") |
| no if | on follow-up fenestrated imaging form, |
| | right renal patent is checked |
| | (FIMG:PATRRA = "PATENT") |
| missing otherwise | |

occlusion, left renal

| yes if | on follow-up fenestrated imaging form, left renal occluded is checked |
|---|---|
| no if | (FIMG:PATLRA = "OCCLUDED") on follow-up fenestrated imaging form, left renal patent is checked (FIMG:PATLRA = "PATENT") |
| missing otherwise | |

occlusion, SMA

| yes if | on follow-up fenestrated imaging form,<br>SMA occluded is checked |
|---|---|
| | (FIMG:PATSMA = "OCCLUDED") |
| no if | on follow-up fenestrated imaging form,<br>SMA patent is checked (FIMG:PATSMA = "PATENT") |
| missing otherwise | |

occlusion, celiac

| ecorasion, conac | |
|-------------------|-----------------------------------------|
| yes if | on follow-up fenestrated imaging form, |
| | celiac occluded is checked |
| | (FIMG:PATCEL = "OCCLUDED") |
| no if | on follow-up fenestrated imaging form, |
| | celiac patent is checked (FIMG:PATCEL = |
| | "PATENT") |
| missing otherwise | |

## 2. Definitions of non-image-related events

At each follow-up visit (each value of FUP:CPEVENT) after the first follow-up visit, each patient is classified as follows:

### creatinine notation:

- C\_b = creatinine on subject history form (LABS:LABCRE)
- C f = creatinine on follow-up form (FUP:LABCRE) at current visit
- C\_p = creatinine on follow-up form (FUP:LABCRE) at previous visit

### creatinine rise

| yes if | $(C_f - C_b) / C_b > 0.30 \text{ AND}$ |
|-------------------|-----------------------------------------|
| | $(C_p - C_b) / C_b > 0.30$ |
| no if | $(C_f - C_b) / C_b \le 0.30 \text{ OR}$ |
| | $(C_p - C_b) / C_b \le 0.30$ |
| missing otherwise | |

## 3. Summary reports for events

At selected visits, the following is reported for each event:

- number of subjects with event = yes
   (number of subjects with event = yes) + (number of subjects with event = no)

The selected visits are as follows:

| • | pre-discharge | (FIMG/FUP:CPEVENT = "PRE_DISCHARGE") |
|---|---------------|--------------------------------------|
| • | 1 month | (FIMG/FUP:CPEVENT = "1 MONTH FUP") |
| • | 6 months | (FIMG/FUP:CPEVENT = "6 MONTH FUP") |
| • | 12 months | (FIMG/FUP:CPEVENT = "12 MONTH FUP") |
| • | 24 months | (FIMG/FUP:CPEVENT = "24 MONTH FUP") |
| • | 36 months | (FIMG/FUP:CPEVENT = "3 YEAR FUP") |
| • | 48 months | (FIMG/FUP:CPEVENT = "4 YEAR FUP") |
| • | other | (FIMG/FUP:CPEVENT = "OTHER") |

## 4. Mortality

### 4.1. General

Each patient will have a follow-up time, defined as follows:

- = months from initial procedure date (PRTH:PROCDT such that PRTH:PROTYP = "INIT IMPLANT") to death date (DTH:DTHDAT), if known to be dead
- = months from initial procedure date (PRTH:PROCDT such that PRTH:PROTYP = "INIT IMPLANT") to last day of reporting period, if not known to be dead

A month will be defined as 30 days.

#### 4.2. All-cause

All-cause mortality will be summarized in the following table:

| | Follow-up time | | | | | | |
|---|---|---|---|---|---|---|---|
| | 1 month | 6 | 12 | 24 | 36 | 48 | 60 |
| | | months | months | months | months | months | months |
| Alive and | | | | | | | |
| in study <sup>a</sup> | | | | | | | |
| Dead to | before | | | | | | |
| date <sup>b</sup> | discharge: <sup>e</sup> | | | | | | |
| | after | | | | | | |
| | discharge:f | | | | | | |
| Censored | | | | | | | |
| to date <sup>c</sup> | | | | | | | |
| Survival | | | | | | | |
| probability <sup>d</sup> | | 2 11 | | | | | |

<sup>&</sup>lt;sup>a</sup>Number of subjects whose follow-up times are greater than the time point.

<sup>&</sup>lt;sup>b</sup>Number of subjects whose follow-up times are less than or equal to the time point and who are known to be dead.

<sup>&</sup>lt;sup>c</sup>Number of subjects whose follow-up times are less than or equal to the time point and who are not known to be dead.

<sup>&</sup>lt;sup>d</sup>The Kaplan-Meier estimate of the survival curve at the time point, with 95-percent confidence interval. The survival curve gives the probability of surviving past a given time.

<sup>&</sup>lt;sup>e</sup>Number of subjects in this cell whose deaths occurred before discharge (PRTH:DSCHDT).

<sup>&</sup>lt;sup>f</sup>Number of subjects in this cell whose deaths occurred after discharge (PRTH:DSCHDT).

## 4.3. AAA-related

Deaths will be classified as AAA-related based on the following definition:

| yes if | death occurs within 30 days of any |
|-------------------|--------------------------------------------|
| yes 11 | • |
| | procedure (initial or secondary) OR |
| | on the death form, "procedure caused or |
| | contributed to death" = yes |
| | (DTH:DTCYNP = "YES" and |
| | DTH:DTHCTX = "PROCEDURE |
| | CAUSED OR CONTRIBUTED TO |
| | DEATH") OR |
| | on the death form, "device caused or |
| | contributed to death" = yes |
| | (DTH:DTCYNP = "YES" and |
| | DTH:DTHCTX = "DEVICE CAUSED OR |
| | CONTRIBUTED TO DEATH") |
| no if | death does not occur within 30 days of any |
| | procedure (initial or secondary) AND |
| | on the death form, "procedure caused or |
| | contributed to death" = no (DTH:DTCYNP |
| | = "NO" and DTH:DTHCTX = |
| | "PROCEDURE CAUSED OR |
| | CONTRIBUTED TO DEATH") AND |
| | on the death form, "device caused or |
| | contributed to death" = no (DTH:DTCYNP |
| | = "NO" and DTH:DTHCTX = "DEVICE |
| | CAUSED OR CONTRIBUTED TO |
| | DEATH") |
| missing otherwise | , |

AAA-related mortality will be summarized in the following table:

| | Follow-up time | | | | | | |
|---|---|---|---|---|---|---|---|
| | 1 month | 6 | 12 | 24 | 36 | 48 | 60 |
| | | months | months | months | months | months | months |
| Alive and | | | | | | | |
| in study <sup>a</sup> | | | | | | | |
| Dead of | before | | | | | | |
| AAA to | discharge: <sup>e</sup> | | | | | | |
| date <sup>b</sup> | after | | | | | | |
| | discharge:f | | | | | | |
| Censored | | | | | | | |
| to date <sup>c</sup> | | | | | | | |
| Survival | | | | | | | |
| probability <sup>d</sup> | | | | | | | |

<sup>a</sup>Number of subjects whose follow-up times are greater than the time point.

<sup>b</sup>Number of subjects whose follow-up times are less than or equal to the time point, who are known to be dead, and whose deaths are AAA-related.

<sup>c</sup>Number of subjects whose follow-up times are less than or equal to the time point and who are not known to be dead, are dead of a cause unrelated to AAA, or are dead of an unknown cause.

<sup>d</sup>The Kaplan-Meier estimate of the survival curve at the time point, with 95-percent confidence interval. The survival curve gives the probability of surviving past a given time.

<sup>e</sup>Number of subjects in this cell whose deaths occurred before initial discharge (PRTH:DSCHDT such that PRTH:PROTYP = "INIT IMPLANT").

<sup>f</sup>Number of subjects in this cell whose deaths occurred after initial discharge (PRTH:DSCHDT such that PRTH:PROTYP = "INIT IMPLANT").

#### 5. Secondary interventions

Each patient will have a follow-up time, defined as follows:

- months from date of initial procedure (PRTH:PROCDT such that PRTH:PROTYP = "INIT IMPLANT") to date of first secondary intervention (PRTH:PROCDT such that PRTH:PROTYP = "ADD ENDO"), if any secondary interventions
- = months from initial procedure date (PRTH:PROCDT such that PRTH:PROTYP = "INIT IMPLANT") to death date (DTH:DTHDAT), if no secondary interventions and known to be dead
- = months from initial procedure date (PRTH:PROCDT such that PRTH:PROTYP = "INIT IMPLANT") to last day of reporting period, if no secondary interventions and not known to be dead

A month will be defined as 30 days.

Secondary interventions will be summarized in the following table:

| | Follow-up time | | | | | | |
|---|---|---|---|---|---|---|---|
| | 1 month | 6 | 12 | 24 | 36 | 48 | 60 |
| | | months | months | months | months | months | months |
| Alive, in | | | | | | | |
| study, and | | | | | | | |
| free of | | | | | | | |
| secondary | | | | | | | |
| interventions <sup>a</sup> | | | | | | | |
| Has | | | | | | | |
| experienced | | | | | | | |
| at least one | | | | | | | |
| secondary | | | | | | | |
| intervention <sup>b</sup> | | | | | | | |
| Censored to | | | | | | | |
| date <sup>c</sup> | | | | | | | |
| Survival | | | | | | | |
| probability <sup>d</sup> | | | | | | | |

<sup>&</sup>lt;sup>a</sup>Number of subjects whose follow-up times are greater than the time point.

<sup>&</sup>lt;sup>b</sup>Number of subjects whose follow-up times are less than or equal to the time point and who experienced at least one secondary intervention.

<sup>&</sup>lt;sup>c</sup>Number of subjects whose follow-up times are less than or equal to the time point and and who have not experienced any secondary interventions.

<sup>&</sup>lt;sup>d</sup>The Kaplan-Meier estimate of the survival curve at the time point, with 95-percent confidence interval. The survival curve gives the probability of surviving past a given time.

#### 6. Validation

A random sample of approximately 5 percent of the subjects will be drawn, and these subjects' data will be audited. Auditing will consist of comparing the data on the remote data capture screens, which are considered source data, to the following derived data sets:

- 1. the web report "patient event report"
- 2. the web report "follow-up time for survival analysis"
- 3. the statistician's working mortality data sets
- 4. the statistician's working secondary intervention data sets

Auditing will be done by people uninvolved in producing the derived data sets.

#### 7. Web reports

#### 7.1. General

All reports are available in Excel or PDF format and can be limited in any of the following ways:

- 1. whether to exclude compassionate use cases (default: do not exclude)
  - a. exclude (CLNO:COMPYN = "NO")
  - b. do not exclude (all cases)
- 2. type of device (default: all subjects):
  - a. fenestrated
    b. visceral
    c. hypogastric
    (PRTH:FORMTP1 = 1)
    (PRTH:FORMTP3 = 1)
- 3. maximum subject number (default: all subjects)
- 4. maximum enrollment date (default: date on which the report is generated), which has the following effects:
  - a. a subject can be included only if his procedure date (PRTH:PROCDT) is less than or equal to the maximum
  - b. a follow-up form can be used only if the visit date (FIMG:APPTDT or FUP:EV DT) is less than or equal to the maximum
  - c. a subject can be counted as dead only if his death date (DTH:DTHDAT) is less than or equal to the maximum
  - d. a secondary intervention can be counted only if the procedure date (PRTH:PROCDT) is less than or equal to the maximum
  - e. the maximum is considered the last day of the reporting period in the definitions of follow-up time in sections 4 and 5

Events are reported at the following visits:

```
pre-discharge
                 (FIMG/FUP:CPEVENT = "PRE_DISCHARGE")
  1 month
                 (FIMG/FUP:CPEVENT = "1 MONTH FUP")
  6 months
                 (FIMG/FUP:CPEVENT = "6 MONTH FUP")
 12 months
                 (FIMG/FUP:CPEVENT = "12 MONTH FUP")
 24 months
                 (FIMG/FUP:CPEVENT = "24 MONTH FUP")
 36 months
                 (FIMG/FUP:CPEVENT = "3 YEAR FUP")
• 48 months
                 (FIMG/FUP:CPEVENT = "4 YEAR FUP")
• other
                 (FIMG/FUP:CPEVENT = "OTHER")
```

# 7.2. Events: Summary report

All events will be included in a single report, which will have one column for each visit and two rows for each event, as follows:

| event | | | visit | |
|------------------|---------------|---------------|---------|--------|
| | | pre-discharge | 1-month | (etc.) |
| endoleak, any | number yes | # | # | |
| | number yes or | # | # | |
| | no | | | |
| endoleak, type I | number yes | # | # | |
| | number yes or | # | # | |
| | no | | | |
| (etc.) | | | | |

### 7.3. Events: Patient-level data set

Each event will have its own report, with one column for each visit and one row for each subject, as follows:

event = endoleak, any

| patient | | visit | |
|---------|---------------|--------------|--------|
| | pre-discharge | 1-month | (etc.) |
| 1 | 0/1/missing | 0/1/ missing | |
| 2 | 0/1/ missing | 0/1/ missing | |
| (etc.) | | _ | |

event = endoleak, type I

| patient | | visit | |
|---------|---------------|--------------|--------|
| | pre-discharge | 1-month | (etc.) |
| 1 | 0/1/ missing | 0/1/ missing | |
| 2 | 0/1/ missing | 0/1/ missing | |
| (etc.) | | _ | |

(etc.)

### 7.4. Mortality and secondary interventions

The summary reports will consist of the tables described in sections 4 and 5. The patient-level reports will have one row for each subject and the following columns:

### Mortality:

- 1. study ID (CLNO:PT)
- 2. Cleveland Clinic ID (CLNO:CLINNO)
- 3. procedure date (PRTH:PROCDT)
- 4. discharge date (PRTH:DSCHDAT)
- 5. date of end of follow-up period, as defined in section 4.1
- 6. length of follow-up period in months, as defined in section 4.1
- 7. indicator of whether subject is dead (0 = no, 1 = yes)
- 8. indicator of whether death is AAA-related, as defined in section 4.3 (0 = no, 1 = yes, NULL = not dead)

### Secondary interventions:

- 1. study ID (CLNO:PT)
- 2. Cleveland Clinic ID (CLNO:CLINNO)
- 3. procedure date (PRTH:PROCDT)
- 4. discharge date (PRTH:DSCHDAT)
- 5. date of end of follow-up period, as defined in section 5
- 6. length of follow-up period in months, as defined in section 5
- 7. indicator of whether subject has had at least one secondary intervention (0 = no, 1 = yes)